CLINICAL TRIAL: NCT07407582
Title: Phase I/II Open Label Trial of Intravenous Sodium Thiosulfate (Pedmark®) as Otoprotectant in Adults Receiving Cisplatin Chemotherapy (STOP-CIS)
Brief Title: Ph. I/II Sodium Thiosulfate for OtoProtection During Cisplatin (STOP-CIS)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Fennec Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006997
Record Dates: First submitted 2026-02-02; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumor Malignancies; Testicular Cancer; Head and Neck Cancer; Thoracic Cancer
Keywords: Cisplatin; Otoprotectant; Cancer; Hearing Impairment; Sodium Thiosulfate; Adults; Solid Tumor
MeSH Terms: conditions — Testicular Neoplasms; Head and Neck Neoplasms; Neoplasms; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Treatment Arm (Experimental): Study participants will receive Pedmark® STS via intravenous infusion after the completion of their standard of care cisplatin infusion.
  Interventions: Drug: Pedmark® STS

INTERVENTIONS:
Drug: Pedmark® STS — Pedmark® STS (20 g/m2) will be given via intravenous infusion over 15-30 minutes, starting 6 hours after the completion of cisplatin infusion. Pedmark® STS will be given each day of cisplatin infusion.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of a drug called Pedmark® sodium thiosulfate (STS) in reducing hearing impairment with standard of care cisplatin therapy. The safety and effectiveness of STS in reducing hearing loss has been well established in children and is approved for use in the pediatric and young adult population. However, information in adult patients is limited. As most cisplatin is administered in the adult population, this investigation would be of benefit.

ELIGIBILITY:
Inclusion Criteria:

* Participants have provided informed consent prior to initiation of any study-specific activities.
* At least 18 years of age, male and female, at the time of signing the informed consent.
* ECOG Performance Status 0-1
* Histologically or cytologically confirmed treatment-naïve cancer.
* Scheduled to receive an FDA-approved, on-label indication, standard of care systemic cisplatin-based regimen (at least 200 mg/m2 cumulative dose) for any untreated any solid malignancy deemed by the treating physician

Exclusion Criteria:

* Prior cisplatin exposure due to a cancer treatment history
* Concurrent ototoxic medication unable to be safely discontinued or switched to a non-toxic alternative
* Planned radiation to the head or neck prior to, during, or within 3 months of completion of cisplatin
* History of severe hypersensitivity to sulfite, sodium thiosulfate, or any components
* Baseline serum sodium > 145 mmol/L or any grade ≥ 3 electrolyte abnormality
* Cisplatin infusion duration greater than 6 hours
* Females during pregnancy or breastfeeding, and childbearing potential, unwilling to use a method of contraception during treatment
* Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment
* Subject likely not to be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (i.e., Clinical Outcome Assessments) to the best of the subject's and investigator's knowledge.
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of intravenous STS to reduce hearing impairment associated with cisplatin | Baseline, after cumulative cisplatin dose (≥ 200 mg/m2), and at 3 months following the conclusion of cisplatin chemotherapy treatment.
  Proportion of participants with Brock grade ≥1 hearing loss determined from audiometry exams. The Brock ototoxicity classification and grading scale are as follows: Grade 0 = hearing threshold less than 40 dB HL at all test frequencies; Grade 1 = hearing threshold greater than or equal to 40 dB HL at 8 kHz only; Grade 2 = hearing threshold greater than or equal to 40 db HL at 4kHz and above; Grade 3 = hearing threshold greater than or equal to 40 dB HL at 2 kHz and above; Grade 4 = hearing threshold greater than or equal to 40 dB HL at 1 kHz and above.

SECONDARY OUTCOMES:
Tolerability of the administration of STS based on the adverse events | At the end of treatment, up to 12 months from baseline.
  Overall safety profile characterized by the type, frequency, severity, duration, and relationship to STS of any adverse events.
Tolerability of the administration of STS: emetic control. | At the end of treatment, up to 12 months from baseline.
  Emetic control (episodes nausea and/or vomiting) will be documented during the clinic visit or hospital stay as per standard practice and assessed using the MASCC Antiemesis Tool (MAT).
Cisplatin pharmacokinetics: area under the plasma concentration versus time curve (AUC) | At the first study treatment visit
  A noncompartmental pharmacokinetic analysis of total and unbound cisplatin will be performed with Phoenix WinNonlin v8.5 (Certara), using a linear method to calculate the area under the plasma concentration versus time curve (AUC) at 4 and 6 hours post-cisplatin dose at the first study treatment visit.
Cisplatin pharmacokinetics: peak plasma concentration (Cmax) | At the first study treatment visit
  A noncompartmental pharmacokinetic analysis of total and unbound cisplatin will be performed with Phoenix WinNonlin v8.5 (Certara), using a linear method to calculate the peak plasma concentration (Cmax) at 4 and 6 hours post-cisplatin dose at the first study treatment visit.
Cisplatin pharmacokinetics: elimination rate constant | At the first study treatment visit
  A noncompartmental pharmacokinetic analysis of total and unbound cisplatin will be performed with Phoenix WinNonlin v8.5 (Certara), using a linear method to calculate the elimination rate constant at 4 and 6 hours post-cisplatin dose at the first study treatment visit.
Cisplatin pharmacokinetics: half-life | At the first study treatment visit
  A noncompartmental pharmacokinetic analysis of total and unbound cisplatin will be performed with Phoenix WinNonlin v8.5 (Certara), using a linear method to calculate the half-life at 4 and 6 hours post-cisplatin dose at the first study treatment visit.
Cisplatin pharmacokinetics: total body clearance | At the first study treatment visit
  A noncompartmental pharmacokinetic analysis of total and unbound cisplatin will be performed with Phoenix WinNonlin v8.5 (Certara), using a linear method to calculate the total body clearance at 4 and 6 hours post-cisplatin dose at the first study treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Davis, PharmD, Study Chair — University of Arizona; Alejandro Recio-Boiles, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No